CLINICAL TRIAL: NCT04287270
Title: Evaluation of Respiratory Muscle Strength in Patients With Multiple System Atrophy
Brief Title: Respiratoy Muscle Strength in Patients With Multiple System Atrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: SAG-B-241018-0566
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2021-03-26 (Actual); Status verified 2021-03

CONDITIONS: Multiple System Atrophy
Keywords: Multiple System Atrophy; Respiratory Muscle Strength; Sniff Nasal Inspiratory Pressure
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Intervention Model Description: Multiple system atrophy patients; Inspiratory muscle strength will be evaluated with sniff nasal inspiratory pressure (SNIP) and maximal inspiratory mouth pressure (PImax). Expiratory muscle strength will be evaluated maximal expiratory mouth pressure (PEmax). Pulmonary function test will be performed.
  Healthy Controls: Inspiratory muscle strength will be evaluated with sniff nasal inspiratory pressure (SNIP) and maximal inspiratory mouth pressure (PImax). Expiratory muscle strength will be evaluated maximal expiratory mouth pressure (PEmax). Pulmonary function test will be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assesment of MSA patients and healthy controls (Other): Demographic information (sex, age, occupation, height, bodyweight ...), clinical and medical status, diagnosis date and Mini-Mental Status Scale data of all participants will be recorded at the first visit. Inspiratory muscle strength will be evaluated with sniff nasal inspiratory pressure and maximal inspiratory mouth pressure, expiratory muscle strength will be evaluated with expiratory mouth pressure. Also, the pulmonary function test will be applied.
  Interventions: Other: Assesment

INTERVENTIONS:
Other: Assesment — Evaluations which explained in the arms section will be made as described.

SUMMARY:
The purpose of this study is; compare respiratory function parameters and respiratory muscle strength in patients with MSA compare to healthy controls, and to evaluate the results of SNIP and PImax in measuring inspiratory muscle strength in MSA patients.

DETAILED DESCRIPTION:
Multiple system atrophy (MSA) is a sporadic, neurodegenerative disease that begins in adulthood, progressive, unexplained. Brain stem degeneration is thought to play a role in respiratory symptoms such as stridor, sleep-related respiratory disturbances and respiratory failure in MSA patients. Respiratory disorders were emphasized and evaluated in MSA during the studies. However, the pattern of pulmonary anomalies or the performance of the inspiratory muscles is not well defined in the MSA.

Inspiratory muscle strength is assessed by voluntary or involuntary tests. The most commonly used reference values are the known maximal inspiratory mouth pressure (PImax) measurement for ease of use. In people with neuromuscular disease, the influence of the orofacial muscles can cause air leakage from the mouth. As a result, low values may be due to air escape which caused by true respiratory muscle weakness, submaximal effort or weakness of the facial muscles.

The purpose of this study is; compare respiratory function parameters and respiratory muscle strength in patients with MSA compare to healthy controls, and to evaluate the results of SNIP and MIP in measuring inspiratory muscle strength in MSA patients.

For this purpose; demographic information (sex, age, occupation, height, body weight ...), clinical and medical status, diagnosis date and Mini Mental Status Scale data of all participants will be recorded at the visit. Inspiratory muscle strength will be evaluated with sniff nasal inspiratory pressure and maximal inspiratory mouth pressure. Expiratory muscle strength will be evaluated with maximal expiratory mouth pressure (PEmax).

ELIGIBILITY:
Inclusion Criteria:

* Being between 40-80 years old
* Have been diagnosed with MSA
* Being under drug treatment
* Being enlightened to participate in the study and filling in the consent form
* Respiratory disease or no history of occupational exposure to affect the respiratory system
* The absence of any physical or mental disability that will prevent the implementation of the tests
* Mini Mental Test score> 24

Exclusion Criteria:

* Any history of neuromuscular disease other than MSA
* Having a diagnosis of psychiatric illness
* Chronic obstructive pulmonary disease (COPD) diagnosis
* The patient is not cooperative
* dementia
* Nasal congestion

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-02-02 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-02-26 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory mouth pressure (PImax) | 15 minutes
  Maximum inspiratory pressure (PImax) is the classic volitional test of inspiratory muscle strength. It is measured as the highest mouth pressure (cmH2O) sustained for 1 s during a maximum inspiratory effort against a quasi occlusion. Evaluation is carried out according to American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria.
Sniff nasal inspiratory pressure (SNIP) | 10 minutes
  Sniff nasal inspiratory pressure (SNIP) measurement is a volitional noninvasive assessment of inspiratory muscle strength. A maximum of 10 sniffs is generally used. It is a simple procedure consisting of measuring peak nasal pressure (cmH2O) as a result of maximal sniff performance through from the end of expiration with the open nostril while the other one is closed.
Maximal expiratory mouth pressure (PEmax) | 15 minutes
  Maximum expiratory pressure (PEmax) is the classic volitional test of expiratory muscle strength. It is measured as the highest mouth pressure (cmH2O) sustained for 1 s during a maximum expiratory effort against a quasi occlusion. Evaluation is carried out according to American Thoracic Society (ATS) / European Respiratory Society (ERS) criteria.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 15 minutes
  Forced vital capacity (FVC) is the volume of air that can forcibly be blown out after full inspiration, measured in liters. FVC is the most basic maneuver in spirometry tests. Pulmonary function test is performed to determine FVC.
Forced expiratory volume in 1 second (FEV1) | 15 minutes
  Forced expiratory volume in 1 second (FEV1) is the volume of air that can forcibly be blown out in first 1 second, after full inspiration. Pulmonary function test is performed to determine FEV1.
FEV1/FVC | 15 minutes
  FEV1/FVC is the ratio of FEV1 to FVC. In healthy adults, this should be approximately 70-80% (declining with age).
Peak expiratory flow (PEF) | 15 minutes
  Peak expiratory flow (PEF) is the maximal flow (or speed) achieved during the maximally forced expiration initiated at full inspiration, measured in liters per minute or in liters per second. Pulmonary function test is performed to determine PEF.

CONTACTS AND LOCATIONS:
Overall Officials: Semra Oguz, PT, PhD, Study Director — Marmara University; Begum Unlu, PT, MSc, Principal Investigator — Marmara University
Locations (1):
- Marmara University Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No